CLINICAL TRIAL: NCT01205282
Title: A Pilot Dose Finding Study of Pioglitazone in Children With ASD
Brief Title: Dose Finding Study of Pioglitazone in Children With Autism Spectrum Disorders (ASD) (PIO)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Evdokia Anagnostou (Individual)
Collaborators: Holland Bloorview Kids Rehabilitation Hospital (Other)
Responsible Party: Sponsor-Investigator, Evdokia Anagnostou, Clinician Scientist, Anagnostou, Evdokia, M.D.
Organization: Anagnostou, Evdokia, M.D. (Individual)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 10-002
Record Dates: First submitted 2010-09-16; First posted 2010-09-20 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2017-03

CONDITIONS: Autism Spectrum Disorders
Keywords: ASD
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pioglitazone (Experimental): A modified dose finding method will be used to determine safety and dose response among three dose levels (0.25mg/kg QD, 0.5mg/kg QD, and 0.75mg/kg QD). There will be 14 weeks of active treatment.
  Interventions: Drug: Pioglitazone
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pioglitazone — A modified dose finding method will be used to determine safety and dose response among three dose levels (0.25mg/kg QD, 0.5mg/kg QD, and 0.75mg/kg QD). The dose has been based on the per weight maximum adult dose. Specifically, the FDA has approved 45mg as the maximum adult dose. For a 60kg adult, this is 0.75mg/kg. There will be 14 weeks of active treatment.
  Arms: Pioglitazone
Drug: Placebo — There will be a 2 week period of placebo run-in.
  Arms: Placebo

SUMMARY:
The investigators propose a pilot, single blind, placebo run-in, dose finding study of pioglitazone in children with autism with the ultimate goal of identifying appropriate dosing and outcome measures for a larger follow-up randomized placebo controlled clinical trial. The specific aims of this study are: 1) To examine the safety of pioglitazone in children with autism spectrum disorders (ASD) ages 5-12 years; 2) To identify appropriate outcome measures to be used in a follow-up multisite randomized control trial of pioglitazone in children with ASD; 3) To determine the maximum tolerated dose to be used in the follow-up multisite randomized controlled trial; 4) To examine the effect of pioglitazone on markers of inflammation (cytokine levels) and oxidative stress (superoxide dismutase, malonyl aldehydes); 5) To explore the relationship between different doses and response to treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female outpatients 5-12 years of age inclusive (see Note below).
2. Meet Diagnostic and Statistical Manual of Mental Disorders, 4th Edition, Text Revision (DSM-IV) criteria. DSM-IV criteria for Autistic Disorder or Asperger's Disorder (autism spectrum disorder) will be confirmed by a clinician with expertise with individuals with ASD. Best estimate Diagnosis will be reached using DSM-IV criteria, the Autism Diagnostic Observation Schedule (ADOS-G) and the Autism Diagnostic Interview-Revised (ADI-R).
3. Have a Clinical Global Impression-Severity (CGI-S) score ≥ 4 (moderately ill) at Baseline.
4. If already receiving stable non-pharmacologic educational, behavioural, and/or dietary interventions, have continuous participation during the preceding 3 months prior to Screening and will not electively initiate new or modify ongoing interventions for the duration of the study.
5. Have normal physical examination and laboratory test results at Screening. If abnormal, the finding(s) must be deemed clinically insignificant by the Investigator.

Exclusion Criteria:

1. Patients born prior to 35 weeks gestational age.
2. Families without sufficient command of the English Language.
3. Patients with any primary psychiatric diagnosis other than autism at Screening.
4. Patients with a current neurological disease, including, but not limited to, movement disorder, tuberous sclerosis, fragile X, and any other known genetic syndromes.
5. Pregnant female patients, female patients who are sexually active, female patients using the birth control pill for whatever reason.
6. Patients with a medical condition that might interfere with the conduct of the study, confound interpretation of the study results, or endanger their own well-being. Patients with evidence or history of malignancy or any significant hematological, endocrine, cardiovascular (including any rhythm disorder), respiratory, renal, hepatic, or gastrointestinal disease. Patients with stable epilepsy (no seizures for 6 months) and on stable doses of antiepileptic medications (no changes in 3 months) will be allowed in the study.
7. Patients taking psychoactive medication(s).
8. Patients taking insulin.
9. Patients unable to tolerate venipuncture procedures for blood sampling.
10. Patients with parent(s)/caregiver(s) who smoke.
11. Patients who have had previous bladder infection(s).
12. Patients with a family history of bladder cancer.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2013-04; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Safety of pioglitazone in children with ASD ages 5-12 years | 16 Weeks
  This will be measured by the Clinical Global Impressions - Improvement Scale - Global (CGI-I-Global)
Safety of pioglitazone in children with ASD ages 5-12 years | 16 Weeks
  This will be measured by the Safety Monitoring Uniform Report Form (SMURF)
Efficacy of outcome measure to be used in a follow-up multisite randomized control trial of pioglitazone in children with ASD | 16 Weeks
  This will be measured by the Aberrant Behavior Checklist (ABC)
Efficacy of outcome measure to be used in a follow-up multisite randomized control trial of pioglitazone in children with ASD | 16 Weeks
  This will be measured the Social Responsiveness Scale (SRS)
Efficacy of outcome measure to be used in a follow-up multisite randomized control trial of pioglitazone in children with ASD | 16 Weeks
  This will be measured by the the Child Yale-Brown Obsessive-Compulsive Scale (CY-BOCS)
Efficacy of outcome measure to be used in a follow-up multisite randomized control trial of pioglitazone in children with ASD | 16 Weeks
  This will be measured by the Repetitive Behavior Scale - Revised (RBS-R)
Efficacy of outcome measure to be used in a follow-up multisite randomized control trial of pioglitazone in children with ASD | 16 Weeks
  This will be measured by the Behavioral Assessment System for Children (BASC-2)
Efficacy of outcome measure to be used in a follow-up multisite randomized control trial of pioglitazone in children with ASD | 16 Weeks
  This will be measured by the Child and Adolescent Symptom Inventory (CASI) - Anxiety Subscale
Maximum tolerated dose to be used in the follow-up multisite randomized controlled trial | 16 Weeks
  Maximum Tolerated Dose (MTD)

SECONDARY OUTCOMES:
Efficacy of pioglitazone on markers of inflammation (cytokine levels) and oxidative stress (superoxide dismutase, malonyl aldehydes) | 16 Weeks
  Cytokine level and oxidative stress marker measurement
Relationship between different doses and response to treatment | 16 Weeks
  Pioglitazone dose and treatment response

CONTACTS AND LOCATIONS:
Overall Officials: Evdokia Anagnostou, M.D., Principal Investigator — Holland Bloorview Kids Rehabilitation Hospital
Locations (1):
- Holland Bloorview Kids Rehabilitation Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Capano L, Dupuis A, Brian J, Mankad D, Genore L, Hastie Adams R, Smile S, Lui T, Odrobina D, Foster JA, Anagnostou E. A pilot dose finding study of pioglitazone in autistic children. Mol Autism. 2018 Nov 26;9:59. doi: 10.1186/s13229-018-0241-5. eCollection 2018. PMID 30498564